CLINICAL TRIAL: NCT00360217
Title: The Efficacy and Short-Term Safety of Docosahexaenoic Acid (DHA) and Statin Therapy for Subjects With Coronary Artery Disease or Cardiac Risk Equivalents With Moderate Hypertriglyceridemia (IIb)
Brief Title: The Triglyceride Lowering Effect of an Omega-3 Fat (DHA) in Addition to Statin Therapy for Patients With CAD or Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maine Center for Lipids and Cardiovascular Health (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2006-08-02; First posted 2006-08-04 (Estimated); Last update posted 2011-11-18 (Estimated); Status verified 2006-07

CONDITIONS: Hypertriglyceridemia (TG>200<500); Hyperlipidemia; Coronary Artery Disease; Coronary Risk Equivalent; Diabetes
Keywords: Omega-3; Triglyceride; Hyperlipidemia; Coronary Artery Disease; Fatty Acids; Safety; Fish Oil; Docosohexanoic Acid
MeSH Terms: conditions — Hypertriglyceridemia; Hyperlipidemias; Coronary Artery Disease; Diabetes Mellitus

INTERVENTIONS:
Drug: docosahexanoic acid (DHA)

SUMMARY:
This study will explore the ability of an algae (ocean plant) omega-3 fat supplement (DHA) to reduce triglyceride levels in patients currently being treated with statin therapy (Zocor or simvastatin, Lipitor or atorvastatin, Pravachol or pravastatin, Crestor or rosuvastatin, etc.) for coronary artery disease(CAD)or risk equivalents (any of the following: heart attack, post angioplasty or stent, post coronary bypass surgery, angina, vascular disease, stroke or diabetes).

The rationale for the study is based around the finding that patients with CAD have an approximately 20 % reduction in the risk of sudden death when treated with fish oil (DHA is one of the ingredients in fish oil). In studies of statin-based therapies, it has been observed that statins reduce the risk of coronary events 20-45%. There has not yet been research trials exploring the combination of the two ingredients (i.e., DHA plus statin) in patient treatment either to reduce recurrent cardiac events or to address another reported finding of fish oils to lower triglyceride levels (triglyceride is a form of "blood fat"). This research project will be a pilot project to assess the safety and effectiveness of DHA "add-on" therapy in patients currently being treated with statins for CAD.

The study hypothesis is to test the effectiveness of DHA as compared to placebo to lower triglyceride levels in the blood. This is a double-blinded randomized clinical trial.

DETAILED DESCRIPTION:
Omega-3 fatty acids (nPUFAs) have been embraced by Expert Panels and Guideline Committees of the American Heart Association as a result of randomized trials documenting reductions in cardiovascular events in patients with coronary artery disease. The antiarrhythmic effect or a modification in the atherogenicity of lipoprotein particles by nPUFA treatment are speculated mechanisms of action. Although precise bioactivity is not clear, nPUFAs have been demonstrated to lower triglyceride (TG) levels. TG reductions have also been demonstrated in three randomized clinical trials where nPUFAs in the form of fish oil containing both eicosapentanoic acid (EPA) and docosahexaenoic acid (DHA) have been added to ongoing statin therapy.

There are at least 8 large randomized clinical trials that have utilized statin agents as monotherapy to reduce cardiovascular events in patients with CAD. These trials have included more than 50,000 patients. The National Cholesterol Education Program (NCEP) recently released a "white paper" further reducing the LDL treatment target to 70 mg% as a result of four recently published trials. Although cardiovascular events rate and mortality reduction of 20-30% have been described, there is still a sizable number of patients experiencing untoward outcomes in spite of ongoing statin therapy. A variety of mechanisms of disease progression have been speculated including ongoing inflammation, insulin resistance and specific species of lipoprotein particles including HDL and LDL sub-classes. There has been recognition by the NCEP that beyond the treatment with statin therapies less tested methods of therapy might need to be applied. These therapies have included the lowering of triglycerides.

It is the purpose of this pilot study to explore the relationship of DHA as a strategy for triglyceride lowering in CAD patients receiving on-going statin therapy and candidates for the yet (untested) recommendation by NCEP of the need to lower triglyceride levels exceeding 200 mg% in statin-treated individuals.

1. This is a single-center, prospective, randomized, double-blinded, placebo-controlled, parallel-group clinical trial of Martek's DHASCO™ versus placebo in subjects with CAD or risk equivalents (including type II DM)
2. There will be a 4-wk run-in period to assure both diet and triglyceride stabilization.
3. After the base-line run-in period, if triglyceride levels exceed 200 mg% they will be eligible to procede with the intervention either placebo or 2 grams of DHA
4. Patients will be treated for an 8 week period. Visits will occur every other week during the treatment cycle.
5. Laboroatory parameters to be followed during the course of the clinical trial includes: beta quantification of lipids, NMR particle analysis of lipoprotein particle size, apoprotein genotyping and other basic chemistry measurements

ELIGIBILITY:
Inclusion Criteria:

* CAD or Risk Equivalent
* On any statin therapy
* At NCEP LDL goal (<100)
* TG>200 mg%

Exclusion Criteria:

* TG>500, TG levels that vary more than 25% during base-line
* Poorly controlled DM
* BMI>40
* Use of fibrates, niacin, other fish oil product

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-01; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Lowering of triglyceride level

SECONDARY OUTCOMES:
Alteration of LDL particle size

CONTACTS AND LOCATIONS:
Overall Officials: Leonard M Keilson, MD, MPH, Principal Investigator — Maine Center for Lipids and Cardiovascular Health
Locations (1):
- Maine Center for Lipids and Cardiovascular Health, Scarborough, Maine, United States